CLINICAL TRIAL: NCT00196586
Title: Pilot Study of Addition of IL-2 to Pegylated Interferon Alpha 2a and Ribavirin for the Treatment of Chronic Hepatitis C in HIV-HCV Coinfected Patients Non Responders to Three Months of Therapy With Pegylated Interferon Alpha 2a and Ribavirin. ANRS HC09 SECOIIA
Brief Title: Efficacy and Safety of Addition of IL-2 to Pegylated Interferon Alpha 2a and Ribavirin in HIV/HCV Coinfected Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Collaborators: Hoffmann-La Roche (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANRS HC09 SECOIIA
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2007-11-16 (Estimated); Status verified 2007-11

CONDITIONS: HIV Infections; Chronic Hepatitis C
Keywords: Chronic Hepatitis C; HIV infection; Interleukin-2; Pegylated interferon alpha 2 a; ribavirin
MeSH Terms: conditions — HIV Infections; Hepatitis C, Chronic | interventions — Interleukin-2; Ribavirin

INTERVENTIONS:
Drug: Interleukin 2
Drug: pegylated interferon alpha 2a
Drug: ribavirin

SUMMARY:
The purpose of this pilot study is to evaluate efficacy and safety of addition of IL-2 to pegylated interferon alpha 2a and ribavirin in HIV-HCV coinfected patients non-responders after three months of standard therapy with pegylated interferon alpha 2a and ribavirin. IL-2 may enhance numbers and function of CD4 T lymphocytes and specific anti-HCV immune responses and could participate to the control of HCV replication

DETAILED DESCRIPTION:
This pilot study evaluate efficacy and safety of addition of IL-2 to pegylated interferon alpha 2a and ribavirin in HIV-HCV coinfected patients non-responders after three months of standard therapy with pegylated interferon alpha 2a and ribavirin Eligible patients should have CD4 cells count higher than 300/mm³ if pretreated by antiretroviral therapy or higher than 400/mm³ if naive of antiretroviral therapy, Metavir score with histological fibrosis score F1, F2 or F3.

Recombinant IL-2 will be given subcutaneously at a dose of 3 MUI twice daily for 5 days every 8 weeks for 5 cycles from week 14 to week 46. This national multicenter study will enroll around 75 patients in order to give IL-2 to 20 non-responders.

The primary endpoint is sustained virologic response, defined by undetectable serum HCV-RNA at week 72, six months after the end of therapy

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection and HCV infection
* Naive of ribavirin
* CD4 higher than 300 if pretreated by antiretroviral therapy or higher than 400 if naive of antiretroviral therapy
* Signed informed consent

Exclusion Criteria:

* Cirrhosis (histological fibrosis score F4 in Metavir score)
* Other liver disease
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75
Dates: Start 2003-04; Study Completion 2006-11

PRIMARY OUTCOMES:
Sustained virologic response, defined by undetectable serum HCV-RNA at week 72, six months after the end of treatment; Safety of IL-2 in combination with pegylated interferon and ribavirin

SECONDARY OUTCOMES:
Virologic response at the end of treatment at week 48, Biochemical response, CD4 cell counts and HIV-RNA plasma levels from baseline to week 72

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Weiss, MD, Principal Investigator — Hopital Européen Georges Pompidou Paris; Jean-Pierre Aboulker, MD, Study Director — Inserm SC10
Locations (1):
- Hopital Européen Georges Pompidou, Paris, France